CLINICAL TRIAL: NCT06805097
Title: Clinical Efficacy of Platelet Transfusion
Acronym: ECLAT
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2025/934
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Thrombocytopaenia; Haematological Malignancies
Keywords: platelet concentrate; transfusion; haemorrhage
MeSH Terms: conditions — Thrombocytopenia; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with severe thrombocytopenia: Patients with haematological malignancies who have severe thrombocytopenia associated with bone marrow failure requiring platelet transfusion and who are able to self-assess bleeding events.
  Interventions: Other: Self-assessment of bleeding events

INTERVENTIONS:
Other: Self-assessment of bleeding events — After each transfusion, the patient completes a daily bleeding event self-assessment (adapted from the WHO bleeding event scale) until the next transfusion or over a period of 10 days.

SUMMARY:
The aim of this study is to analyze the effect of the storage time of platelet concentrates on the occurrence of bleeding events during prophylactic platelet transfusions in patients with hematological malignancies.

DETAILED DESCRIPTION:
Since 2017, the preparation processes and shelf life of platelet concentrates (PCs) have been changed to increase transfusion safety and optimise transfusion processes. These changes have led to an increase in the total number of PCs transfused, a decrease in the number of platelets per PC and an increase in the number of platelets transfused per patient. Previous studies have shown that longer storage of platelets contributes to less in vivo recirculation of transfused platelets. Studies of haemostatic efficacy have generally not reported a significant effect. However, the haemostatic efficacy of PC stored for more or less than 5 days has not been evaluated. The ECLAT multicentre prognostic cohort study will prospectively and comparatively evaluate the haemorrhagic event in haematology patients with severe thrombocytopenia transfused according to the duration of PC storage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with haematological malignancies or bone marrow aplasia with severe thrombocytopenia due to bone marrow failure related to the disease or treatments received
* Severe thrombocytopenia requiring transfusion
* Patient able to self-assess bleeding events
* Non-opposition of the subject to participate in the study
* Registered with the French social security system or benefiting from such a system.

Exclusion Criteria:

* Acute promyelocytic leukaemia
* Curative dosage of anticoagulants
* Treatment with antiplatelet agents
* Patient with proven thrombocytopenia of immunological origin, or disseminated intravascular coagulation
* Patients with a clinically significant haemorrhagic event (WHO grade 2) in the 48 hours prior to transfusion
* Indication for deplasmatised, cryopreserved and reduced-volume PCs
* Patient refusing transfusion of labile blood products
* Pregnant women or breast-feeding mothers
* Adults subject to a legal protection measure or unable to express their consent
* Persons deprived of their liberty by a judicial or administrative decision; persons under compulsory psychiatric care; persons admitted to a health or social care institution for purposes other than research
* Subject in the exclusion period of another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for haematological malignancy with severe thrombocytopenia associated with bone marrow failure and requiring platelet transfusion
Sampling Method: Non-Probability Sample
Enrollment: 343 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Grade 2 or higher bleeding event | 7 days
  Grade 2 or higher bleeding event, depending on platelet shelf life.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: Undecided